CLINICAL TRIAL: NCT02420340
Title: Using The HOPES Program in Transition Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Glencliff Home (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 27956
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Serious Mental Illness; Psychosocial Rehabilitation
Keywords: Serious Mental Illness; Psychosocial Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HOPES Group (Other): Participants will participate in twice weekly sessions of the HOPES program until curriculum is completed (approximately 1 year) or discharge from Glencliff home
  Interventions: Behavioral: HOPES Program ("Helping Older People Experience Success")

INTERVENTIONS:
Behavioral: HOPES Program ("Helping Older People Experience Success") — Weekly group skills training classes aimed at improving skills and knowledge in areas related to successful living in the community including: independent living, healthy living, social skills, leisure skills, and management of health care.

SUMMARY:
This pilot study will collect information about the the potential to use an evidence-based skills training program designed for older people with serious mental illness (SMI), the Helping Older People Experience Success (HOPES) program, to help nursing home residents with SMI gain the skills needed to successfully live in the community.

DETAILED DESCRIPTION:
This pilot study will collect information about the the potential to use an evidence-based skills training program designed for older people with serious mental illness (SMI), the Helping Older People Experience Success (HOPES) program, to help nursing home residents with SMI gain the skills needed to successfully live in the community. Although HOPES was originally designed to help older people with SMI maintain their residence in the community, the curriculum holds promise for helping nursing home residents with SMI to learn how to return to life in the community. Positive findings would be used to develop a grant application for a larger study of HOPES in nursing home residents with SMI. To evaluate the feasibility and acceptability of HOPES in nursing home settings, the investigators will enroll up to 12 residents of the Glencliff Home in Glencliff, New Hampshire. Participants will be individuals interested in discharge from Glencliff and are willing to attend multiple weekly skills training classes and several assessment sessions. Study participation will last until 6 months after discharge from Glencliff.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder as defined in participants' chart
* An expressed willingness to be discharged from Glencliff Home to the community.
* Voluntary informed consent for participation in the study by the participant or by the participant's legally designated guardian

Exclusion Criteria:

* Terminal physical illness OR significant medical instability
* Inability to speak or and understand English
* Primary or co-morbid diagnosis of dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Attendence-70% attendance or higher of HOPES groups over the course of the intervention | 12 months
  attendance records
Change in Functional Skills (University California San Diego Performance-Based Skills Assessment) | Baseline, 12 months, 6 month follow-up
  University California San Diego Performance-Based Skills Assessment

SECONDARY OUTCOMES:
Change in Medication Adherence and Management (Medication Management Ability Assessment) | Baseline, 12 months, 6 month follow-up
  Medication Management Ability Assessment
Change in Social Skills (Social Skills Performance Assessment) | Baeline, 12 months, 6 month follow-up
  Social Skills Performance Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Glencliff Home, Glencliff, New Hampshire, United States

REFERENCES:
- [Result] Mueser KT, Pratt SI, Bartels SJ, Swain K, Forester B, Cather C, Feldman J. Randomized trial of social rehabilitation and integrated health care for older people with severe mental illness. J Consult Clin Psychol. 2010 Aug;78(4):561-73. doi: 10.1037/a0019629. PMID 20658812